CLINICAL TRIAL: NCT03257345
Title: VEST: The UK Vedolizumab Real Life Experience Study in Inflammatory Bowel Disease
Acronym: VEST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other); Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Principal Investigator, Fraser Cummings, Consultant Gastroenterologist, University Hospital Southampton NHS Foundation Trust
Other Study IDs: RHM MED1307
Record Dates: First submitted 2017-08-17; First posted 2017-08-22 (Actual); Last update posted 2018-09-21 (Actual); Status verified 2018-09

CONDITIONS: Ulcerative Colitis; Crohn's Disease
Keywords: Real world outcomes
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

SUMMARY:
Vedolizumab has been approved for the treatment of both ulcerative colitis and Crohn's disease. The aim of this study is to capture the early real life UK experience of vedolizumab including the outcomes of treatment, describing the patient population treated, drug persistence, IBD control PROM, durable remission, tolerance and safety.

ELIGIBILITY:
Inclusion Criteria:

* Participants being given vedolizumab as part of routine care, and vedo naïve prior to study
* Age 18 or over
* Written informed consent obtained from patient for participation in the UK IBD Registry

Exclusion Criteria:

* Patient unwilling to take part in the UK IBD Registry
* Unable to obtain written informed consent
* Patient is, in the opinion of the investigator, not suitable to participate in the study
* Patients with contraindications to the use of vedolizumab

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with inflammatory bowel disease due to start vedolizumab for the first time as part of routine therapy.
Sampling Method: Probability Sample
Enrollment: 360 (Estimated)
Dates: Start 2017-02-03 (Actual); Primary Completion 2019-09-30 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Steroid-free remission | Week 56
  Steroid-free remission at one year as defined by an HBI at week 56 of ≤4 or a UCDAI of ≤2

SECONDARY OUTCOMES:
Remission and response | Multiple
  Remission and response rates at week 6, 14, 30 and 54
Durable remission | Multiple
  Durable remission / response i.e. at week 14, 30 and 54
Effect of vedolizumab | TBC
  Effect of vedolizumab on disease activity as measured by the PRO2, IBD Control PROM, Physician's Global Assessment and biomarkers of disease activity
HES data | 1 year
  Healthcare usage at 1 year using HES data
Tolerance and safety | 1 year
  Tolerance and safety of vedolizumab at 1 year
Description of disease | TBC
  Description of the demographics, disease phenotype, disease and treatment history and concomitant medication use of patients receiving vedolizumab

CONTACTS AND LOCATIONS:
Locations (22):
- United Kingdom (22):
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - Royal Devon and Exeter NHS Foundation Trust, Exeter, Devon
  - Brighton and Sussex University Hospitals NHS Trust, Brighton, East Sussex
  - Kingston Hospital NHS Foundation Trust, Kingston, Greater London
  - Barts Health NHS Trust, London, Greater London
  - London North West Healthcare NHS Trust, London, Greater London
  - University College London Hospitals NHS Foundation Trust, London, Greater London
  - Guy's and St Thomas' NHS Foundation Trust, London, Greater London
  - King's College Hospital NHS Foundation Trust, London, Greater London
  - University Hospital Southampton NHS Foundation Trust, Southampton, Hampshire
  - West Hertfordshire Hospitals NHS Trust, Watford, Hertfordshire
  - Maidstone and Tunbridge Wells NHS Foundation Trust, Maidstone, Kent
  - United Lincolnshire Hospitals NHS Trust, Grantham, Lincolnshire
  - Aintree University Hospital NHS Foundation Trust, Liverpool, Merseyside
  - York Teaching Hospital NHS Foundation Trust, York, North Yorkshire
  - Shrewsbury and Telford Hospital NHS Trust, Shrewsbury, Shropshire
  - Barnsley Hospital NHS Foundation Trust, Barnsley, South Yorkshire
  - Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire
  - West Suffolk NHS Foundation Trust, Bury St Edmunds, Suffolk
  - The Newcastle upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear
  - The Royal Wolverhampton NHS Trust, Wolverhampton, West Midlands
  - Calderdale and Huddersfield NHS Foundation Trust, Huddersfield, West Yorkshire